CLINICAL TRIAL: NCT05709028
Title: Fosfomycin Versus Standard of Care in Children With Antibiotic-resistant Urinary Tract Infections: A Non-inferiority, Pragmatic, Multi-centre Adaptive Trial to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of Oral Fosfomycin in Children With Antibiotic-resistant Urinary Tract Infections.
Brief Title: Fosfomycin Versus Standard of Care in Children With Antibiotic-resistant Urinary Tract Infections
Acronym: FosUTI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FosUTI
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with an intervention arm and an active control arm (standard-of care)
Masking Description: Open-label study. Statisticians will be blind to groups when analysing results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral fosfomycin (Experimental): * Children who have been diagnosed with an uncomplicated UTI will be administered a single dose of oral fosfomycin trometamol. Then, on Day 2 either;
    1. Stop if the child has clinically improved, or
    2. Give a second dose of oral fosfomycin trometamol if the child has ongoing fever or clinical symptoms consistent with an uncomplicated UTI, or
    3. Give an additional 8 days of oral fosfomycin trometamol with repeat doses every 48 hours (to make up a total 10-day treatment duration) if the child has evidence of a complicated UTI.
  * Children who have been diagnosed with a complicated UTI will be administered repeat doses of oral fosfomycin trometamol every 48 hours until the child has received a total 10-day course of antibiotics with presumed or proven efficacy against the urinary pathogen.
  Interventions: Drug: Fosfomycin
- Standard of Care antibiotics (Active Comparator): * Children who have been diagnosed with an uncomplicated UTI will be administered a 3-day course of standard of care (SOC) antibiotics with known efficacy against the urinary pathogen. Then, on Day 3 either;
    1. Stop of the child has clinically improved, or
    2. Give an additional 48 hours of SOC antibiotics if the child has ongoing fever or clinical symptoms consistent with an uncomplicated UTI, or
    3. Give an additional 7 days of SOC antibiotics (to make up a total 10-day duration) if the child has evidence of a complicated UTI.
  * Children who have been diagnosed with a complicated UTI will be administered a total 10-day course of SOC antibiotics with known efficacy against the urinary pathogen.
  Interventions: Drug: Standard of care antibiotics

INTERVENTIONS:
Drug: Fosfomycin — Fosfomycin trometamol is a white crystalline powder which is very soluble in water. The granules are mixed with 90ml of cool water for the constitution to dissolve and will be administered soon after reconstitution. Each 30ml will contain 1g fosfomycin base.
  * Children ≥ 6 months to <1 year old will be administered 30ml (=1g fosfomycin base) of dissolved solution and the remainder discarded for each dose.
  * Children ≥ 1 to 11 years will be administered 60ml (=2g fosfomycin base) of dissolved solution and the remainder discarded for each dose.
  * Children ≥12 and <18 years will be administered the entire 90ml solution (= 3g fosfomycin base) for each dose.
  Arms: Oral fosfomycin
Drug: Standard of care antibiotics — Standard of care antibiotics will be chosen by the treating clinician according to institutional prescribing practices, local antibiograms and medication availability.
  Arms: Standard of Care antibiotics

SUMMARY:
Urinary tract infections (UTIs) are among the most common bacterial infections in children. Up to 50% of UTI's are caused by multi-drug resistant ESBL-producing gram negative bacteria that do not respond to treatment with oral penicillin's or cephalosporins. Instead, children often require hospital admission to receive broad-spectrum intravenous antibiotics when they may otherwise be safely managed at home; resulting in prolonged hospital stays and an increased use of health resources. Fosfomycin is a broad-spectrum antibiotic discovered in 1969 that remains susceptible to a large number of organisms due to its low international use. Fosfomycin can be prepared as an oral solution with an orange/tangerine flavour and is currently approved for use in females >12 years old. Despite extensive evidence of its efficacy in adults and safety in neonates, the use of fosfomycin in children remains limited and fosfomycin is not currently licensed for use in children <12 years old in Australia.

The aim of this clinical trial is to compare the use of oral fosfomycin against standard of care antibiotics for the treatment of antibiotic resistant urinary tract infections in children. The main questions the trial aims to answer are:

1. Is oral fosfomycin non-inferior in efficacy to the current standard of care for the treatment of antibiotic-resistant urinary tract infections in children?
2. Is oral fosfomycin a safe and well-tolerated antibiotic in children?
3. What is the best dosing regimen of oral fosfomycin for the treatment of antibiotic-resistant UTIs in children?

DETAILED DESCRIPTION:
This is a Phase 3, non-inferior, pragmatic, multi-centre, adaptive, randomised clinical trial.

Up to 300 participants aged ≥6 months to <18 years of age with a clinical and microbiological diagnosis of an antibiotic-resistant urinary tract infection will be recruited for the trial. Children will be randomised 1:1 to receive either oral fosfomycin (the intervention) or standard of care. The duration of antibiotic treatment will be dependent on whether the child's UTI is complicated or uncomplicated. Children with at least two of the following signs and symptoms will meet criteria of having a complicated UTI: fever, nausea or vomiting, other signs or symptoms of systemic illness: including chilld or rigors, significant fatigue, irritability or malaise above baseline, flank or back pain, ultrasound findings suggestive of an upper renal tract infection, a known history of structural and/or mechanical urological abnormalities, patients with a stent in situ or known renal tract calculi, patients who are immunocompromised. Children who do not meet the criteria for a 'complicated' UTI will meet criteria for an 'uncomplicated' UTI.

For children allocated to the standard of care (S)C) arm: the choice of antibiotic will be as per physician preference based on institutional prescribing practices, local antibiograms and medication availability. Children with an uncomplicated UTI will be prescribed a 3-day course of SOC antibiotics. Then, on Day 3 either; (a) Stop if the child has clinically improved, or (b) Give an additional 48 hours of SOC antibiotics if the child has ongoing fever or clinical symptoms consistent with an uncomplicated UTI, or (c) Give an additional 7 days of SOC antibiotics (to make up a total 10-day duration) if the child has evidence of a complicated UTI. Children with a complicated UTI diagnosis at the time of enrolment will be administered a total 10-day course of SOC antibiotics.

For children allocated to the intervention arm: Children with an uncomplicated UTI will be administered a single dose of oral fosfomycin trometamol. Then, on Day 2 either; (a) Stop if the child has clinically improved, or (b) Give an additional dose of oral fosfomycin trometamol if the child has ongoing fever or clinical symptoms consistent with an uncomplicated UTI, or (c) Give an additional 8 days of oral fosfomycin trometamol with repeat doses every 48 hours (to make up a total 10-day treatment duration) if the child has evidence of a complicated UTI. Children with a complicated UTI diagnosis at the time of enrolment will be administered a total 10-day course of oral fosfomycin trometamol with repeat doses administered every 48 hours.

Children enrolled into the oral fosfomycin group as well as children enrolled in the standard of care group who receive an oral antibiotic will be asked to complete a tolerability questionnaire following the first dose of the oral antibiotic. The child's parent and a member of their clinical team will also complete this questionnaire. All examinations, investigations and clinical interventions during the study period will be tailored to the child's needs as per routine standard of care. Clinical observations and results will be recorded on a case report form and entered into a secure electronic database. At Day 3, 10 and 28 after enrolment, parents will receive an SMS questionnaire to monitor their ongoing health, capture adverse events and/or capture their medication adherence.

50 children aged ≥6 months to <12 who have been randomised to the fosfomycin arm will be co-enrolled in a pharmacokinetic sub-study. For these children, two blood samples will be taken within 24 hours after the first dose of fosfomycin to determine the plasma fosfomycin concentrations. Co-enrolment into the pharmacokinetic sub-study is optional and will only be performed at a subset of study sites.

ELIGIBILITY:
Inclusion Criteria:

Children aged ≥6 months to <18 years with:

1. Symptoms consistent with a clinical diagnosis of a UTI (as per the treating clinician); AND
2. Microbiological confirmation: Defined as a urine culture revealing a predominant growth of a bacterial uropathogen [≥10^6 CFU/L, or ≥10^3 CFU/mL] together with ≥10x10^6 white blood cells on microscopy; AND
3. The bacterial uropathogen is a non-pseudomonal gram-negative organism likely to cause urinary tract infections in children; being one of either: Escherichia coli, Proteus spp., Klebsiella spp., Enterobacter spp., Serratia spp., or Citrobacter spp., AND
4. The uropathogen has in vitro evidence of resistance to all oral penicillins and oral first- and second- generation cephalosporins (or is presumed to be resistant based on the pattern of phenotypic testing); AND
5. The patient has not yet received >48 hours of antibiotics with in vitro activity against the urinary pathogen prior to enrolment.

   Exclusion Criteria:
6. Evidence of bacteraemia due to the same uropathogen within the same clinical illness; OR
7. Evidence of infection at a secondary site (such as meningitis or endocarditis); OR
8. Children with features suggestive of sepsis (defined as requiring inotropic support, or >20ml/kg fluid bolus); OR
9. Children who are unable to tolerate or absorb oral antibiotics; OR
10. Children with severe renal unsifficiency (creatinine clearance <10ml/minute/1.73m^2); OR
11. Known allergy to fosfomycin; OR
12. A decision by the primary treating physician that enrolment in the trial is not in the child's best interest.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Treatment failure within 28 days after enrolment between patients treated with standard of care versus oral fosfomycin. | 28 days
  Treatment failure is defined as:
  1. Persistent or recurrent (clinical and microbiologically-confirmed) diagnosis of a UTI between 7 and 28 days after enrolment, with the same uropathogen; or
  2. Decision to switch to an alternative antibiotic due to perceived treatment failure; or
  3. Isolation of the same pathogenic organism from a new sterile site between 7 and 28 days after enrolment;

SECONDARY OUTCOMES:
Occurrence of treatment-related adverse events to Day 28 | 28 days
Occurrence of serious adverse events attributable to UTI to Day 28 | 28 days
Evidence of primary treatment failure, defined as: a) Persistent fever (>38.0C) attributable to UTI at 72h after enrolment; and/or b) Failure to return to baseline health at 28 days after enrolment | 28 days
Evaluation of the cost of hospital resources in the first 28 days of enrolment in children receiving standard of care versus oral fosfomycin; including: a) Cost of prescribed drugs b) Cost of hospital services (inpatient and outpatient) | 28 days
Assessment of the tolerability of oral antibiotic therapy in children, using a 5-point facial hedonic scale immediately after the first oral dose | Day 1
  To assess the tolerability of oral fosfomycin, children ≥3 years will be asked immediately after administration of their first dose of fosfomycin or alternative oral antibiotic (if prescribed within SOC), to record how much he or she liked the sample by putting a mark on a 5-point facial hedonic scale (ranging from 1, dislike very much; to 5, liked very much); and whether they would be happy to take the medication again if required. The parent and treating nurse or doctor will also be asked independently to give a score, using separate 5-point hedonic scales, based on their perception of how the child reacted to the taste of oral fosfomycin or alternative oral antibiotic.

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe Williams, Principal Investigator — University of Sydney
Locations (5):
- Australia (5):
  - Sydney Childrens Hospital, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Royal Childrens Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No
Efficacy and AEs/SAEs will be summarised and pooled. Deidentified individual data will be shared with the DSMB and ethics for SAEs only.
  Investigators have the protocols and the ICFs. SAP will be available for all investigators once authored. Reports and analytical code will be shared when approved by trial statisticians.